CLINICAL TRIAL: NCT01599481
Title: Effectiveness and Cost Effectiveness of Individual Career Management for People With Anxiety and Depression: A Randomised Controlled Trial
Brief Title: Career Management to Improve Education, Employment and Retention for People With Anxiety and Depression
Acronym: CAREER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Claire Price, Employment & Social Inclusion Manager, South London and Maudsley NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SLAM-ICM-1011
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Anxiety; Depression
Keywords: Common mental illness; Supported Employment; Anxiety; Depression; Sickness absence
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Employment, Supported; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Standard Care (IAPT Therapy) + Individual Career Management (ICM)
  Interventions: Behavioral: Individual Career Management (ICM); Behavioral: Standard Care
- Control (Active Comparator): Standard Care (IAPT Therapy)
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Individual Career Management (ICM) — The intervention will be Individual Career Management (ICM) support for a six month period. ICM consists of individually tailored support to help an individual to obtain and retain in employment. ICM follows the seven principles of supported employment (often referred to an Individual Placement and Support), but includes the additional principles of career counselling, motivational coaching, education and training support, and specialist job retention support. The length and frequency of ICM support sessions is determined by the needs of the client.
  Other Names: IPS; Supported Employment
  Arms: Intervention
Behavioral: Standard Care — A package of psychological therapy delivered by an Improving Access to Psychological Therapies (IAPT) practitioner.
  Other Names: IAPT; CBT

SUMMARY:
The aim of the investigation is to evaluate the effectiveness and costeffectiveness of a model of supported employment (the Individual Career Management (ICM) model) designed to help people with common mental illness return to work.

DETAILED DESCRIPTION:
The design of the study is a randomised controlled trial of two groups in a natural setting (intervention group vs control group). The primary outcome is paid employment. Standard care for all participants is a package of psychological therapy (IAPT). The intervention is an additional package of employment support (ICM) delivered alongside standard care.

The intervention group and control group will both receive standard care. The intervention group will receive ICM support in addition to standard care and the control group will be given details of other employment programmes in the local area, in line with current IAPT practice. The control period will last six months. There will be no fewer than 184 participants in the study (92 in each arm).

The study will take place at the Southwark Psychological Therapies Service at the SLaM NHS Foundation Trust. Patients that meet the inclusion criteria will be invited to attend an interview where written informed consent and baseline measures will be obtained. The participant will then be randomly assigned to either the intervention or control group. All participants will be invited to attend a second interview at the end of a six month period where followup measures will be taken. If the intervention is available at this time, control group participants may then be offered the opportunity to receive it.

A randomised controlled trial of supported employment for people with common mental health problems has never been carried out in the UK, therefore this study will be the first of its kind. The results will help to determine if ICM is an effective and costeffective service and will provide the foundations for further research in this area.

ELIGIBILITY:
Inclusion Criteria:

* Must be either unemployed or off sick for at least two weeks if employed at the time of entry to the study
* Must be legally allowed to work in the UK
* Must be between the age of 18-65 for men, and 18-60 for women (based on UK retirement age)
* Must have received an IAPT assessment and been offered psychological therapy
* Must not have been receiving therapy for more than one month
* Must be interested in obtaining competitive employment
* Must have given full written consent to participate in the study

Exclusion criteria:

* People who are employed and attending work or off sick for less than two weeks at the time of entry to the study
* People who do not have the legal right to work in the UK
* People who have not yet received an IAPT assessment
* People who have received an IAPT assessment but not eligible for psychological therapy
* People who have been receiving therapy for more than one month
* People who are not interested in obtaining competitive employment
* People who do not give written consent or who lack mental capacity to give consent at the time of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Length of Competitive Employment | 6 months
  Length of competitive employment during the 6 month study period. The following definition of competitive employment will be used:
  1. A job paying at least the national minimum wage.
  2. A job located in a mainstream setting not set aside for people with disabilities.
  3. A job that is not owned by the ICM service.

SECONDARY OUTCOMES:
Working Hours | 6 months
  Average number of hours worked each week
Time to Employment | 6 months
  Number of days between baseline date and the employment start date.
Salary | 6 months
  Average weekly salary over the 6 month period
Number of Jobs | 6 months
  Number of different jobs held during the 6 month period
Job Terminations | 6 months
  Number of job terminations over the 6 month period and the reason for each termination
Other occupational activity | 6 months
  Non-competitive employment (e.g. sheltered work), education, training or volunteering
Anxiety | 6 months
  Generalised Anxiety Disorder Assessment (GAD 7) score
Depression | 6 months
  Patient Health Questionnaire (PHQ-9) score
Social Functioning | 6 months
  Work and Social Adjustment Scale (WSAS)
Health-related quality of Life | 6 months
  EQ-5D score
Work-related quality of Life | 6 months
  WRQoL score
Self Esteem | 6 months
  Rosenberg Self Esteem Scale
Career Search Efficacy | 6 months
  Career Search Efficacy Scale (CSES) score
Return to Work Efficacy | 6 months
  Return to Work Self Efficacy Scale (RTW-SE) score
Productivity | 6 months
  Absenteeism and presenteeism questions from the World Health Organization's Health and Work Performance Questionnaire (HPQ)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Price, CPsychol, Principal Investigator — South London and Maudsley NHS Foundation Trust
Locations (1):
- Southwark Psychological Therapies Service, London, United Kingdom